CLINICAL TRIAL: NCT06187493
Title: Efficacy of ACEi Versus SGLT2i in the Treatment of Patients With Diabetic Kidney Disease : Head to Head RCT
Brief Title: Treatment of Patients With Diabetic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ismael ahmed amin mohammed alaraby, Director of the Health Affairs Directorate, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: diabetic kidney
Record Dates: First submitted 2023-12-06; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Kidney Disease
Keywords: Efficacy of ACEi versus SGLT2i
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Lisinopril; Enalapril; dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of ACEi (Other): Patients receive an ACEi medication, such as lisinopril, enalapril, or ramipril. These drugs work by blocking the production of angiotensin II, a hormone that can constrict blood vessels and raise blood pressure.
  Interventions: Drug: lisinopril, enalapril
- Efficacy of SGLT2i (Other): Patients receive an SGLT2i medication, such as dapagliflozin, empagliflozin, or canagliflozin. These drugs work by preventing the kidneys from reabsorbing glucose from the urine, leading to lower blood sugar levels and potentially reducing the risk of kidney damage.
  Interventions: Drug: dapagliflozin, empagliflozin

INTERVENTIONS:
Drug: lisinopril, enalapril — 1. Both arms should aim to achieve optimal blood pressure control, typically defined as a systolic blood pressure below 130 mmHg and a diastolic blood pressure below 80 mmHg. This can be achieved through lifestyle modifications, additional medications, or a combination of both.
  2. Maintaining good glycemic control is also important for both arms. This can be achieved through diet, exercise, and diabetes medications.
  3. Both arms may also receive other supportive care measures for DKD, such as protein restriction, dietary counseling, and management of other co-morbidities like anemia and hyperlipidemia.
  Arms: Efficacy of ACEi
Drug: dapagliflozin, empagliflozin — 1. Both arms should aim to achieve optimal blood pressure control, typically defined as a systolic blood pressure below 130 mmHg and a diastolic blood pressure below 80 mmHg. This can be achieved through lifestyle modifications, additional medications, or a combination of both.
  2. Maintaining good glycemic control is also important for both arms. This can be achieved through diet, exercise, and diabetes medications.
  3. Both arms may also receive other supportive care measures for DKD, such as protein restriction, dietary counseling, and management of other co-morbidities like anemia and hyperlipidemia.
  Arms: Efficacy of SGLT2i

SUMMARY:
Due to irrespective of the limitations associated with estimated glomerular filtration rate (eGFR), it is crucial to develop new treatments that can effectively address these concerns. So, this study aimed to compare the effectiveness of SGlT2i versus ACEi in the progression of diabetic kidney disease including progression of albuminuria. Doubling of serum creatinine and need for renal replacement therapy

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is the leading cause of end stage renal disease (ESRD) worldwide and continues to be the major contributor to kidney replacement therapy (KRT).

Despite the significant decline in diabetes-related complications in recent decades, the same trend cannot be observed in chronic kidney disease (CKD) patients due to DKD that requires KRT. Hence, there exists a significant requirement for novel treatment approaches that can enhance glycemic control while minimizing the risk of hypoglycemia, as well as reducing cardiovascular and renal risks within this population. Irrespective of the limitations associated with estimated glomerular filtration rate (eGFR), it is crucial to develop new treatments that can effectively address these concerns.

ACE inhibitors may delay the progression of nephropathy and reduce the risks of cardiovascular events in hypertensive patients with diabetes mellitus type I and type II.

SGLT2i have become the new standard of care for slowing CKD progression in patients with type 2 diabetes mellitus (T2DM, due to their specific renal and cardiovascular protective effects that are independent of the main metabolic and glucose-lowering effects.

Research questions:

Q1. Is there a significant effect of ACEi in treatment of patients with diabetic kidney disease.

Q2: Is there is a significant effect of SGLT2i in treatment of patients with diabetic kidney disease.

Q3: Which is more significantly efficient in treatment of patients with diabetic kidney disease (ACEi versus SGLT2i)

ELIGIBILITY:
Inclusion Criteria:

* Patients that suffer from Diabetic kidney disease (DKD)

Exclusion Criteria:

* Genital mycotic infections
* Urosepsis and Pyelonephritis
* Lower limb amputation
* diabetic Ketoacidosis
* Euglycemic DKA
* Acute Kidney Injury
* Hypoglycemia
* Fournier Gangrene
* Hypersensitivity Reactions
* Bone fracture
* Bladder cancer
* Hyperkalemia
* Dyslipidemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
prevention of the development of DKD and alter its natural progression. | baseline≥3 months-year
  Primary Outcome:
  Time to development of DKD: Measured as the time from randomization to the first occurrence of any of the following events:
  Sustained (≥3 months) albumin-to-creatinine ratio (UACR) ≥300 mg/g End-stage kidney disease (ESKD) requiring dialysis or kidney transplantation
  Measurement Tools:
  UACR: Measured in urine samples using commercial laboratory assays. eGFR: Estimated using creatinine levels and demographic data through formulas like CKD-EPI.
  Cardiovascular events and mortality: Ascertained through medical records and national death registries.
  Unit of Measure:
  Time to DKD development: Years or months Change in UACR: mg/g eGFR decline: mL/min/1.73 m² per year Cardiovascular events and mortality: Incidence per 70patient-years

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Tohamy, prof, Study Director — Assiut University; Walaa khalifa, prof, Study Director — Assiut University